CLINICAL TRIAL: NCT05965011
Title: Walking on 'Four Legs' to Manage Falls and Fear of Falling
Brief Title: Nordic Walking to Manage Falls and Fear of Falling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Mohammad Auais, PhD (Other)
Responsible Party: Sponsor-Investigator, Dr. Mohammad Auais, PhD, Assistant Professor, School Of Rehabilitation Therapy, Queen's University
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 6030812
Record Dates: First submitted 2023-06-15; First posted 2023-07-28 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Risk of Falling
Keywords: Fear of Falling; Nordic Walking; Older adults
MeSH Terms: interventions — Exercise; Nordic Walking

STUDY DESIGN:
Intervention Model Description: This study will be a pilot trial conducted as a two-arm, parallel, single-blind, randomized controlled trial.
Who Masked: Outcomes Assessor
Masking Description: The single-blind design will involve that the assessors are unaware of the group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Nordic walking) (Experimental): Nordic walking training. These coaching principles will focus on highlighting the participants' strengths and resourcefulness, setting goals, and utilizing solution-focused problem-solving techniques to achieve those goals during practice and related activities . This group sessions will be conducted biweekly to ensure appropriate progression and adherence to the guidelines set by the International Nordic Walking Federation.
  In addition to the supervised group sessions, participants will also receive supervised NW training from a certified NW instructor. Participants will be encouraged to set goals and develop strategies to facilitate independent practice for at least three 30-minute sessions per week over a period of 10 weeks. These unsupervised sessions aim to encourage participants to engage in regular practice outside of the group sessions.
  Interventions: Other: Exercise training
- Control (phone calls) (No Intervention): The control group will receive regular contact to control for attention and maintain participant engagement throughout the study. Over the course of the 10 weeks, participants in this group will receive 5 biweekly phone calls from the study's graduate research assistant (RA).
  During each phone call, the RA will engage in discussions with participants about leading a healthy lifestyle in general, covering topics such as proper nutrition and adequate sleep. Additionally, the RA will gather safety-related data, including information on any falls that may have occurred. The phone calls will also serve as reminders for participants about upcoming assessments and their importance in the study. The investigators will provide a training session to the control group following the completion of the study if they are interested.

INTERVENTIONS:
Other: Exercise training — The intervention will be a combination of both supervised and unsupervised sessions. Participants in the Nordic Walking (NW) treatment group will attend 5 one-hour group sessions, which will incorporate coaching principles.
  Other Names: Nordic walking
  Arms: Intervention (Nordic walking)

SUMMARY:
This is a pilot study that aims to test the feasibility and safety of a novel Nordic Walking (NW) activity program for community-dwelling older adults who are at risk of falling or experience fear of falling (FOF). The study also aims to determine the distribution and effect sizes of outcomes to inform future sample size calculations and explore participants' perspectives of the intervention.

Participants will be asked to:

* Attend training sessions to learn proper Nordic Walking techniques.
* Engage in supervised Nordic Walking sessions for a specified duration and frequency.
* Keep a log of their walking activities and any falls or near falls experienced.
* Complete questionnaires to assess their fear of falling and overall physical activity levels.

If there is a comparison group:

Researchers will compare the intervention group, consisting of older adults participating in the Nordic Walking program, with a control group of older adults who do not receive the intervention. The comparison will be made to determine if Nordic Walking has a significant impact on reducing falls and fear of falling compared to the control group.

DETAILED DESCRIPTION:
Introduction:

this is a pilot study that aims to test the feasibility and safety of a novel Nordic Walking (NW) activity program for community-dwelling older adults who are at risk of falling or experience fear of falling (FOF). The study also aims to determine the distribution and effect sizes of outcomes to inform future sample size calculations and explore participants' perspectives of the intervention.

Background:

Falls and fear of falling are significant concerns among older adults, leading to physical impairments, psychological trauma, and a decline in abilities and quality of life. Exercise has been shown to be effective in improving muscle strength, balance, mobility, and postural control, all of which are risk factors for falls and FOF. However, traditional exercise programs have limitations in terms of cost, sustainability, and long-term adherence. Nordic Walking, a low-risk and low-tech intervention, has emerged as a promising alternative, offering numerous physical and mental health benefits.

Study Design:

The study will be conducted in two stages. Stage One will involve a two-arm, parallel, single-blind, randomized controlled pilot trial. Forty older adults at risk of falling will be recruited and randomly assigned to either a 10-week NW intervention group or a control group. The intervention group will receive supervised NW training sessions and will be coached to practice independently. The control group will receive regular phone calls to discuss healthy lifestyle habits.

Outcome Measures:

The study will collect feasibility and safety data, including recruitment, adherence, and follow-up rates, as well as adverse events. Effectiveness outcomes will be assessed using measures such as the Timed Up and Go (TUG) test, Stay Independent Falls Risk Assessment Tool, Falls Efficacy Scale-International (FES-I), Activities-Specific Balance Confidence Scale, and the Four-Square Step Test (FSST).

Data Analysis:

Descriptive statistics will be used to characterize participants and feasibility measures. Hedge's effect size and confidence intervals will be calculated. Independent samples t-tests and chi-square tests will be used to compare the intervention and control groups. The main focus of the analysis will be to estimate the effect size, test the intervention's feasibility and safety, and inform future studies.

Sample Size:

The study aims to recruit 40 participants (20 per group) to ensure study robustness and account for potential dropouts.

Stage Two:

In the second stage, qualitative interviews will be conducted with all participants in the intervention group to gather feedback on the acceptability, perceived value, barriers, and facilitators of participating. The data will be analyzed using interpretive description to identify themes and categories.

ELIGIBILITY:
Inclusion Criteria:

* Must be 60+ years old.
* Be at risk of falling, as determined by the Stay Independent Falls Risk Assessment Tool. This validated tool is recommended by the STEADI fall prevention program to evaluate risk of falling.

Exclusion Criteria:

* Inability to use walking poles due to medical conditions.
* Inability to walk 400m independently.
* Having a medical condition such as unstable cardiorespiratory status, impending angioplasty, or ataxia/dyskinesia (unsteady, staggering gait) that prevents them from participating in physical activities or using walking poles is prohibited.
* Taking part in any other structured exercise program.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Estimate the effect size of intervention (Cohen's D) | Through study completion, an average of 1.5 years
  Effect size estimation is vital in assessing the impact of interventions like Nordic walking and planning future studies. It involves quantifying the magnitude of the intervention's effect on the outcome variable.
Evaluate the adherence rate to the intervention (as a measure of feasibility) | Through study completion, an average of 1.5 years
  Participant Adherence to the Intervention: This measure examines the extent to which participants adhere to the prescribed Nordic walking program. It involves tracking the frequency, duration, and intensity of Nordic walking sessions completed by participants. Adherence rates can be calculated based on the number of sessions attended or completed as planned.
Assess safety of the intervention | Through study completion, an average of 1.5 years
  Monitoring Adverse Events: We systematically record and monitor any adverse events or incidents during the study. This includes injuries, discomfort, or any negative effects reported by participants.

SECONDARY OUTCOMES:
Timed Up and Go (TUG) to assess fall risk | Pre (week 0) /post intervention (week 11)
  The Timed Up and Go (TUG) test is a widely used clinical assessment tool to evaluate mobility and functional mobility, specifically in older adults. While it is not specifically designed to determine the risk of falling, it can provide valuable information that is correlated with fall risk. The TUG test measures the time it takes for an individual to stand up from a chair, walk a set distance (typically 3 meters), turn around, return to the chair, and sit down again.
Fear of Falling: Fear of falling will be measured by the Falls Efficacy Scale-International (FES-I) | Pre (week 0) /post intervention (week 11)
  Scale: Falls Efficacy Scale-International (FES-I) Minimum Value: 0 (not at all confident) Maximum Value: 100 (completely confident) Interpretation: In the FES-I, higher scores indicate greater fear of falling. Therefore, a higher score on the FES-I reflects a worse outcome, indicating a higher level of fear and reduced confidence in performing daily activities without falling. Conversely, a lower score on the FES-I suggests a better outcome, indicating a lower level of fear and greater confidence in performing activities without fear of falling.
Performance on the Four-Square Step Test (FSST) will be measured to assess balance. | Pre (week 0) /post intervention (week 11)
  The Four-Square Step Test (FSST) does not yield a specific score on a scale like some other assessments. Instead, the FSST primarily focuses on the time taken to complete the test and the occurrence of errors or missteps.
  When assessing FSST performance, the following information is typically recorded:
  Completion Time: The time the individual takes to complete the FSST is measured in seconds. A shorter completion time generally indicates better balance and agility.
  Errors or Missteps: The number of errors or missteps made by the individual during the FSST is recorded. Errors can include stepping outside the designated squares, incorrect foot placement, or loss of balance. Fewer errors suggest better balance control and coordination.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Rehabilitation Therapy, Queens University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hughes VA, Frontera WR, Wood M, Evans WJ, Dallal GE, Roubenoff R, Fiatarone Singh MA. Longitudinal muscle strength changes in older adults: influence of muscle mass, physical activity, and health. J Gerontol A Biol Sci Med Sci. 2001 May;56(5):B209-17. doi: 10.1093/gerona/56.5.b209. PMID 11320101
- [Background] Krasovsky T, Banina MC, Hacmon R, Feldman AG, Lamontagne A, Levin MF. Stability of gait and interlimb coordination in older adults. J Neurophysiol. 2012 May;107(9):2560-9. doi: 10.1152/jn.00950.2011. Epub 2012 Feb 1. PMID 22298827
- [Background] Herman T, Giladi N, Gurevich T, Hausdorff JM. Gait instability and fractal dynamics of older adults with a "cautious" gait: why do certain older adults walk fearfully? Gait Posture. 2005 Feb;21(2):178-85. doi: 10.1016/j.gaitpost.2004.01.014. PMID 15639397
- [Background] Beauchet O, Annweiler C, Allali G, Berrut G, Herrmann FR, Dubost V. Recurrent falls and dual task-related decrease in walking speed: is there a relationship? J Am Geriatr Soc. 2008 Jul;56(7):1265-9. doi: 10.1111/j.1532-5415.2008.01766.x. Epub 2008 May 26. PMID 18510582
- [Background] Bertera EM, Bertera RL. Fear of falling and activity avoidance in a national sample of older adults in the United States. Health Soc Work. 2008 Feb;33(1):54-62. doi: 10.1093/hsw/33.1.54. PMID 18326450
- [Background] Keast M-L. Nordic walking: introducing a new low-impact exercise system for cardiac rehabilitation patients. Minto prevention and rehabilitation center, University of Ottawa Heart Institute. 2009:13- 14.
- [Background] Ossowski Z, Wawryniku M, Česnaitiene V. Influence of nordic walking training on static and dynamic body balance among the elderly. Baltic Journal of Health and Physical Activity. 2015;7(1):72-80.
- [Background] Karawan A, Porcari J, Butta H, Postmus A, Stoughton L, Larkin J. Effects of 12 weeks of walking or exerstriding on upper body strength and endurance. Medicine & Science in Sports & Exercise. 1992;24(5):S138.
- [Background] Kortas J, Kuchta A, Prusik K, Prusik K, Ziemann E, Labudda S, Cwiklinska A, Wieczorek E, Jankowski M, Antosiewicz J. Nordic walking training attenuation of oxidative stress in association with a drop in body iron stores in elderly women. Biogerontology. 2017 Aug;18(4):517-524. doi: 10.1007/s10522-017-9681-0. Epub 2017 Feb 22. PMID 28229255
- [Background] Dalton C, Nantel J. Nordic Walking Improves Postural Alignment and Leads to a More Normal Gait Pattern Following Weeks of Training: A Pilot Study. J Aging Phys Act. 2016 Oct;24(4):575-582. doi: 10.1123/japa.2015-0204. Epub 2016 Aug 24. PMID 27051072
- [Background] Willson J, Torry MR, Decker MJ, Kernozek T, Steadman JR. Effects of walking poles on lower extremity gait mechanics. Med Sci Sports Exerc. 2001 Jan;33(1):142-7. doi: 10.1097/00005768-200101000-00021. PMID 11194099
- [Background] Reelick MF, van Iersel MB, Kessels RP, Rikkert MG. The influence of fear of falling on gait and balance in older people. Age Ageing. 2009 Jul;38(4):435-40. doi: 10.1093/ageing/afp066. Epub 2009 May 18. PMID 19451658
- [Background] Rubenstein LZ, Vivrette R, Harker JO, Stevens JA, Kramer BJ. Validating an evidence-based, self-rated fall risk questionnaire (FRQ) for older adults. J Safety Res. 2011 Dec;42(6):493-9. doi: 10.1016/j.jsr.2011.08.006. Epub 2011 Nov 17. PMID 22152267
- [Background] Stevens JA. The STEADI Tool Kit: A Fall Prevention Resource for Health Care Providers. IHS Prim Care Provid. 2013 Sep;39(9):162-166. No abstract available. PMID 26766893
- [Background] van Zyl LE, Roll LC, Stander MW, Richter S. Positive Psychological Coaching Definitions and Models: A Systematic Literature Review. Front Psychol. 2020 May 6;11:793. doi: 10.3389/fpsyg.2020.00793. eCollection 2020. PMID 32435218
- [Background] International Nordic Walking Federation. http://inwa-nordicwalking.com/. Accessed May 2021.
- [Background] Bullo V, Gobbo S, Vendramin B, Duregon F, Cugusi L, Di Blasio A, Bocalini DS, Zaccaria M, Bergamin M, Ermolao A. Nordic Walking Can Be Incorporated in the Exercise Prescription to Increase Aerobic Capacity, Strength, and Quality of Life for Elderly: A Systematic Review and Meta-Analysis. Rejuvenation Res. 2018 Apr;21(2):141-161. doi: 10.1089/rej.2017.1921. Epub 2017 Nov 20. PMID 28756746
- [Background] Shumway-Cook A, Brauer S, Woollacott M. Predicting the probability for falls in community-dwelling older adults using the Timed Up & Go Test. Phys Ther. 2000 Sep;80(9):896-903. PMID 10960937
- [Background] Delbaere K, Close JC, Mikolaizak AS, Sachdev PS, Brodaty H, Lord SR. The Falls Efficacy Scale International (FES-I). A comprehensive longitudinal validation study. Age Ageing. 2010 Mar;39(2):210-6. doi: 10.1093/ageing/afp225. Epub 2010 Jan 8. PMID 20061508
- [Background] Powell LE, Myers AM. The Activities-specific Balance Confidence (ABC) Scale. J Gerontol A Biol Sci Med Sci. 1995 Jan;50A(1):M28-34. doi: 10.1093/gerona/50a.1.m28. PMID 7814786
- [Background] Dite W, Temple VA. A clinical test of stepping and change of direction to identify multiple falling older adults. Arch Phys Med Rehabil. 2002 Nov;83(11):1566-71. doi: 10.1053/apmr.2002.35469. PMID 12422327
- [Background] Sullivan GM, Feinn R. Using Effect Size-or Why the P Value Is Not Enough. J Grad Med Educ. 2012 Sep;4(3):279-82. doi: 10.4300/JGME-D-12-00156.1. No abstract available. PMID 23997866
- [Background] Mangione KK, Craik RL, Palombaro KM, Tomlinson SS, Hofmann MT. Home-based leg-strengthening exercise improves function 1 year after hip fracture: a randomized controlled study. J Am Geriatr Soc. 2010 Oct;58(10):1911-7. doi: 10.1111/j.1532-5415.2010.03076.x. PMID 20929467
- [Background] Moore CG, Carter RE, Nietert PJ, Stewart PW. Recommendations for planning pilot studies in clinical and translational research. Clin Transl Sci. 2011 Oct;4(5):332-7. doi: 10.1111/j.1752-8062.2011.00347.x. PMID 22029804
- [Background] Julious SA. Sample size of 12 per group rule of thumb for a pilot study. Pharmaceutical Statistics: The Journal of Applied Statistics in the Pharmaceutical Industry. 2005;4(4):287-291.
- [Background] Thorne S, Kirkham SR, MacDonald-Emes J. Interpretive description: a noncategorical qualitative alternative for developing nursing knowledge. Res Nurs Health. 1997 Apr;20(2):169-77. doi: 10.1002/(sici)1098-240x(199704)20:23.0.co;2-i. PMID 9100747
- [Background] Soriano TA, DeCherrie LV, Thomas DC. Falls in the community-dwelling older adult: a review for primary-care providers. Clin Interv Aging. 2007;2(4):545-54. doi: 10.2147/cia.s1080. PMID 18225454
- [Background] Parachute. Fall prevention. 2014. https://parachute.ca/en/injury-topic/fall-prevention-for-seniors/. Accessed Mar 2021
- [Background] Falls: Assessment and Prevention of Falls in Older People. London: National Institute for Health and Care Excellence (NICE); 2013 Jun. Available from http://www.ncbi.nlm.nih.gov/books/NBK258885/ PMID 25506960
- [Background] Tinetti ME, Powell L. Fear of falling and low self-efficacy: a case of dependence in elderly persons. J Gerontol. 1993 Sep;48 Spec No:35-8. doi: 10.1093/geronj/48.special_issue.35. No abstract available. PMID 8409238
- [Background] Mane AB, Sanjana T, Patil PR, Sriniwas T. Prevalence and correlates of fear of falling among elderly population in urban area of Karnataka, India. J Midlife Health. 2014 Jul;5(3):150-5. doi: 10.4103/0976-7800.141224. PMID 25317002
- [Background] Tinetti ME, Richman D, Powell L. Falls efficacy as a measure of fear of falling. J Gerontol. 1990 Nov;45(6):P239-43. doi: 10.1093/geronj/45.6.p239. PMID 2229948
- [Background] Murphy SL, Dubin JA, Gill TM. The development of fear of falling among community-living older women: predisposing factors and subsequent fall events. J Gerontol A Biol Sci Med Sci. 2003 Oct;58(10):M943-7. doi: 10.1093/gerona/58.10.m943. PMID 14570863
- [Background] Auais M, French S, Alvarado B, Pirkle C, Belanger E, Guralnik J. Fear of Falling Predicts Incidence of Functional Disability 2 Years Later: A Perspective From an International Cohort Study. J Gerontol A Biol Sci Med Sci. 2018 Aug 10;73(9):1212-1215. doi: 10.1093/gerona/glx237. PMID 29220420
- [Background] Parker SG, Corner L, Laing K, Nestor G, Craig D, Collerton J, Frith J, Roberts HC, Sayer AA, Allan LM, Robinson L, Cowan K; multiple conditions in later life priority setting partnership. Priorities for research in multiple conditions in later life (multi-morbidity): findings from a James Lind Alliance Priority Setting Partnership. Age Ageing. 2019 May 1;48(3):401-406. doi: 10.1093/ageing/afz014. PMID 30892604
- [Background] Rimer J, Dwan K, Lawlor DA, Greig CA, McMurdo M, Morley W, Mead GE. Exercise for depression. Cochrane Database Syst Rev. 2012 Jul 11;(7):CD004366. doi: 10.1002/14651858.CD004366.pub5. PMID 22786489
- [Background] Bula CJ, Monod S, Hoskovec C, Rochat S. Interventions aiming at balance confidence improvement in older adults: an updated review. Gerontology. 2011;57(3):276-86. doi: 10.1159/000322241. Epub 2010 Oct 29. PMID 21042008
- [Background] Howe TE, Rochester L, Neil F, Skelton DA, Ballinger C. Exercise for improving balance in older people. Cochrane Database Syst Rev. 2011 Nov 9;2011(11):CD004963. doi: 10.1002/14651858.CD004963.pub3. PMID 22071817
- [Background] Huang TT, Yang LH, Liu CY. Reducing the fear of falling among community-dwelling elderly adults through cognitive-behavioural strategies and intense Tai Chi exercise: a randomized controlled trial. J Adv Nurs. 2011 May;67(5):961-71. doi: 10.1111/j.1365-2648.2010.05553.x. Epub 2011 Jan 7. PMID 21214623
- [Background] Watzek D, Mischler E, Sonam D, et al. Effectiveness and economic evaluation of therapeutic nordic walking in patients with psychosomatic disorders: A pragmatic randomized controlled trial. Psychology. 2016;6(11):665-675.
- [Background] Finnegan S, Bruce J, Skelton DA, Withers EJ, Lamb SE; PreFIT Study Group. Development and delivery of an exercise programme for falls prevention: the Prevention of Falls Injury Trial (PreFIT). Physiotherapy. 2018 Mar;104(1):72-79. doi: 10.1016/j.physio.2017.06.004. Epub 2017 Jun 27. PMID 28801033
- [Background] Thompson PD, Arena R, Riebe D, Pescatello LS; American College of Sports Medicine. ACSM's new preparticipation health screening recommendations from ACSM's guidelines for exercise testing and prescription, ninth edition. Curr Sports Med Rep. 2013 Jul-Aug;12(4):215-7. doi: 10.1249/JSR.0b013e31829a68cf. No abstract available. PMID 23851406
- [Background] Yamauchi T, Islam MM, Koizumi D, Rogers ME, Rogers NL, Takeshima N. Effect of home-based well-rounded exercise in community-dwelling older adults. J Sports Sci Med. 2005 Dec 1;4(4):563-71. eCollection 2005 Dec. PMID 24501569
- [Background] Dishman RK. Increasing and maintaining exercise and physical activity. Behavior Therapy. 1991;22(3):345-378. 10
- [Background] Cyarto EV, Brown WJ, Marshall AL. Retention, adherence and compliance: important considerations for home- and group-based resistance training programs for older adults. J Sci Med Sport. 2006 Oct;9(5):402-12. doi: 10.1016/j.jsams.2006.06.020. Epub 2006 Sep 5. PMID 16911871
- [Background] Yan T, Wilber KH, Simmons WJ. Motivating high-risk older adults to exercise: does coaching matter? Home Health Care Serv Q. 2011 Apr;30(2):84-95. doi: 10.1080/01621424.2011.569670. PMID 21590567
- [Background] Church TS, Earnest CP, Morss GM. Field testing of physiological responses associated with Nordic Walking. Res Q Exerc Sport. 2002 Sep;73(3):296-300. doi: 10.1080/02701367.2002.10609023. PMID 12230336
- [Background] Jordan AN, Olson TP, Earnest CP, Morss GM, Church TS. Metabolic cost of high intensity poling while nordic walking versus normal walking. Medicine & Science in Sports & Exercise. 2001;33(5):S86.
- [Background] Figard-Fabre H, Fabre N, Leonardi A, Schena F. Physiological and perceptual responses to Nordic walking in obese middle-aged women in comparison with the normal walk. Eur J Appl Physiol. 2010 Apr;108(6):1141-51. doi: 10.1007/s00421-009-1315-z. Epub 2009 Dec 20. PMID 20091181
- [Background] Mikalacki M, Cokorilo N, Katic R. Effect of nordic walking on functional ability and blood pressure in elderly women. Coll Antropol. 2011 Sep;35(3):889-94. PMID 22053573
- [Background] Bulinska K, Kropielnicka K, Jasinski T, Wojcieszczyk-Latos J, Pilch U, Dabrowska G, Skorkowska-Telichowska K, Kalka D, Zywar K, Paszkowski R, Wozniewski M, Szuba A, Jasinski R. Nordic pole walking improves walking capacity in patients with intermittent claudication: a randomized controlled trial. Disabil Rehabil. 2016;38(13):1318-24. doi: 10.3109/09638288.2015.1077398. Epub 2015 Aug 25. PMID 26305413
- [Background] Breyer MK, Breyer-Kohansal R, Funk GC, Dornhofer N, Spruit MA, Wouters EF, Burghuber OC, Hartl S. Nordic walking improves daily physical activities in COPD: a randomised controlled trial. Respir Res. 2010 Aug 22;11(1):112. doi: 10.1186/1465-9921-11-112. PMID 20727209
- [Background] van Eijkeren FJ, Reijmers RS, Kleinveld MJ, Minten A, Bruggen JP, Bloem BR. Nordic walking improves mobility in Parkinson's disease. Mov Disord. 2008 Nov 15;23(15):2239-43. doi: 10.1002/mds.22293. PMID 18816697
- [Background] Reuter I, Mehnert S, Leone P, Kaps M, Oechsner M, Engelhardt M. Effects of a flexibility and relaxation programme, walking, and nordic walking on Parkinson's disease. J Aging Res. 2011;2011:232473. doi: 10.4061/2011/232473. Epub 2011 Mar 30. PMID 21603199
- [Background] Ossowski ZM, Skrobot W, Aschenbrenner P, Cesnaitiene VJ, Smaruj M. Effects of short-term Nordic walking training on sarcopenia-related parameters in women with low bone mass: a preliminary study. Clin Interv Aging. 2016 Nov 30;11:1763-1771. doi: 10.2147/CIA.S118995. eCollection 2016. PMID 27942207
- [Background] Morso L, Hartvigsen J, Puggaard L, Manniche C. Nordic walking and chronic low back pain: design of a randomized clinical trial. BMC Musculoskelet Disord. 2006 Oct 2;7:77. doi: 10.1186/1471-2474-7-77. PMID 17014731
- [Background] Sanchez-Lastra MA, Torres J, Martinez-Lemos I, Ayan C. Nordic walking for women with breast cancer: A systematic review. Eur J Cancer Care (Engl). 2019 Nov;28(6):e13130. doi: 10.1111/ecc.13130. Epub 2019 Aug 6. PMID 31389108
- [Background] Gomenuka NA, Oliveira HB, Silva ES, Costa RR, Kanitz AC, Liedtke GV, Schuch FB, Peyre-Tartaruga LA. Effects of Nordic walking training on quality of life, balance and functional mobility in elderly: A randomized clinical trial. PLoS One. 2019 Jan 30;14(1):e0211472. doi: 10.1371/journal.pone.0211472. eCollection 2019. PMID 30699211
- [Background] Mannerkorpi K, Nordeman L, Cider A, Jonsson G. Does moderate-to-high intensity Nordic walking improve functional capacity and pain in fibromyalgia? A prospective randomized controlled trial. Arthritis Res Ther. 2010;12(5):R189. doi: 10.1186/ar3159. Epub 2010 Oct 13. PMID 20942911
- [Background] Suija K, Pechter U, Kalda R, Tahepold H, Maaroos J, Maaroos HI. Physical activity of depressed patients and their motivation to exercise: Nordic Walking in family practice. Int J Rehabil Res. 2009 Jun;32(2):132-8. doi: 10.1097/MRR.0b013e32831e44ef. PMID 19065108
- [Background] Ossowski Z, Prusik K, Prusik K, Kortas J, Wiech M. Nordic walking training and physical fitness in elderly women. Polish Journal of Sport and Tourism. 2015;21(4):253-257.
- [Background] Parkatti T, Perttunen J, Wacker P. Improvements in functional capacity from Nordic walking: a randomized-controlled trial among elderly people. J Aging Phys Act. 2012 Jan;20(1):93-105. doi: 10.1123/japa.20.1.93. Epub 2011 Sep 15. PMID 21949243
- [Background] Šokelienė V, Česnaitienė VJ. The influence of nordic walking on physical fitness of elderly people. Baltic Journal of Sport and Health Sciences. 2011;3(82).
- [Background] Ben Mansour K, Gorce P, Rezzoug N. The impact of Nordic walking training on the gait of the elderly. J Sports Sci. 2018 Oct;36(20):2368-2374. doi: 10.1080/02640414.2018.1458396. Epub 2018 Mar 27. PMID 29582714
- [Background] Gomenuka NA, Oliveira HB, da Silva ES, Passos-Monteiro E, da Rosa RG, Carvalho AR, Costa RR, Rodriguez Paz MC, Pellegrini B, Peyre-Tartaruga LA. Nordic walking training in elderly, a randomized clinical trial. Part II: Biomechanical and metabolic adaptations. Sports Med Open. 2020 Jan 13;6(1):3. doi: 10.1186/s40798-019-0228-6. PMID 31932999
- [Background] Lee HS, Park JH. Effects of Nordic walking on physical functions and depression in frail people aged 70 years and above. J Phys Ther Sci. 2015 Aug;27(8):2453-6. doi: 10.1589/jpts.27.2453. Epub 2015 Aug 21. PMID 26357424
- [Background] Gmiat A, Jaworska J, Micielska K, Kortas J, Prusik K, Prusik K, Lipowski M, Radulska A, Szupryczynska N, Antosiewicz J, Ziemann E. Improvement of cognitive functions in response to a regular Nordic walking training in elderly women - A change dependent on the training experience. Exp Gerontol. 2018 Apr;104:105-112. doi: 10.1016/j.exger.2018.02.006. Epub 2018 Feb 9. PMID 29432893
- [Background] Chalmers I, Glasziou P. Avoidable waste in the production and reporting of research evidence. Lancet. 2009 Jul 4;374(9683):86-9. doi: 10.1016/S0140-6736(09)60329-9. Epub 2009 Jun 12. No abstract available. PMID 19525005
- [Background] Meisner BA, Boscart V, Gaudreau P, Stolee P, Ebert P, Heyer M, Kadowaki L, Kelly C, Levasseur M, Massie AS, Menec V, Middleton L, Sheiban Taucar L, Thornton WL, Tong C, van den Hoonaard DK, Wilson K. Interdisciplinary and Collaborative Approaches Needed to Determine Impact of COVID-19 on Older Adults and Aging: CAG/ACG and CJA/RCV Joint Statement. Can J Aging. 2020 Sep;39(3):333-343. doi: 10.1017/S0714980820000203. Epub 2020 Jun 10. PMID 32408910
- [Background] Schrack JA, Wanigatunga AA, Juraschek SP. After the COVID-19 Pandemic: The Next Wave of Health Challenges for Older Adults. J Gerontol A Biol Sci Med Sci. 2020 Sep 16;75(9):e121-e122. doi: 10.1093/gerona/glaa102. No abstract available. PMID 32315025
- [Background] Cunningham C, O' Sullivan R, Caserotti P, Tully MA. Consequences of physical inactivity in older adults: A systematic review of reviews and meta-analyses. Scand J Med Sci Sports. 2020 May;30(5):816-827. doi: 10.1111/sms.13616. Epub 2020 Feb 4. PMID 32020713
- [Background] Santini ZI, Jose PE, York Cornwell E, Koyanagi A, Nielsen L, Hinrichsen C, Meilstrup C, Madsen KR, Koushede V. Social disconnectedness, perceived isolation, and symptoms of depression and anxiety among older Americans (NSHAP): a longitudinal mediation analysis. Lancet Public Health. 2020 Jan;5(1):e62-e70. doi: 10.1016/S2468-2667(19)30230-0. PMID 31910981
- [Background] Queens Gazette. How the School of Rehabilitation Therapy is breaking down barriers to physiotherapy in the Kingston community. In. Kingston, Ontraio, Canada 2021:https://healthsci.queensu.ca/stories/feature/how-school-rehabilitation-therapy-breaking-down barriers-physiotherapy-kingston.
- [Background] Steffen TM, Hacker TA, Mollinger L. Age- and gender-related test performance in community-dwelling elderly people: Six-Minute Walk Test, Berg Balance Scale, Timed Up & Go Test, and gait speeds. Phys Ther. 2002 Feb;82(2):128-37. doi: 10.1093/ptj/82.2.128. PMID 11856064
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Yardley L, Beyer N, Hauer K, Kempen G, Piot-Ziegler C, Todd C. Development and initial validation of the Falls Efficacy Scale-International (FES-I). Age Ageing. 2005 Nov;34(6):614-9. doi: 10.1093/ageing/afi196. PMID 16267188